CLINICAL TRIAL: NCT06844617
Title: A Trial of the Difference in Staff Time Involved in Repositioning Proned Patients in the ICU Using the 'BathMat' Compared With Standard Care
Brief Title: A Trial of Staff Time With Proned Patients in the ICU Using the 'BathMat'
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal United Hospitals Bath NHS Foundation Trust (Other)
Collaborators: University of Bath (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 333769
Record Dates: First submitted 2025-02-05; First posted 2025-02-25 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-01

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS); Proning; Intensive Care Medicine
Keywords: BathMat; Proning; Proned; Repositioning; Intensive Care; ICU; ITU; Bath Mat
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: This is a randomised, multicentre, single blind crossover study of repositioning in ventilated proned patients in ICU using the BathMat vs conventional care.
Who Masked: Participant
Masking Description: Participants will be unconscious and unaware of which arm they are involved in. Due to the nature of the device, blinding of care providers or investigators is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Repositioning using standard care (No Intervention): Patients are repositioned while proned using standard care on each unit, every 2-4 hours.
- Repositioning using BathMat (Experimental): Patients are repositioned using the BathMat, every 2-4 hours.
  Interventions: Device: BathMat

INTERVENTIONS:
Device: BathMat — Repositioning patients using the BathMat
  Arms: Repositioning using BathMat

SUMMARY:
Proning is a way of helping people who are very sick and have trouble breathing. It involves lying patients on their front to get more oxygen into their body. This process happens in a part of the hospital called the Intensive Care Unit, and can last up to 16 hours per day.

When in this position, doctors need to turn the patients' head and move their arms every 2-4 hours. Doctors call this repositioning. It helps prevent sores as well as other injuries. To do this, the health care team slide the patient up the bed, so that their (supported) head hangs over the end of the mattress. The head is then turned before the patient is slid back down the bed; their arms are then moved into a different position. This is currently performed by a team of 5+ staff and takes lots of time and resources. The process is also potentially dangerous because it requires a lot of movement which can hurt patients or staff.

To make repositioning easier and safer, a group of doctors and engineers have created a new device. It is like a cushion that goes under the patient and inflates. This allows staff to reposition patients without needing to slide the patient on the bed. This also reduces the number of staff needed and lowers the risk to patients and staff. Feedback from staff, patients and the public are being used to help improve the system.

To see if the new device works well in other hospitals, the investigators are planning to do a study with 30 patients in up to 4 different hospitals. This will last 14 months, and they will collect information on how well it performs. They will ask patients if they want to take part and will collect feedback after they leave hospital. During the study, staff from each hospital will monitor the device to make sure it is safe and record how useful it is. Any problems will be recorded, and staff will be asked for their opinions on how it affects their work. As well as monitoring safety, they will record the time saving achieved. This is important as it allows repositioning more often, which may reduce pressure sores. It also allows staff to spend more time focusing on other patients and important tasks. To share the results with other doctors, the researchers will write reports and give presentations. If successful, they will start making and selling the device to help sick patients on Intensive Care.

DETAILED DESCRIPTION:
Approximately 235,000 patients per year are admitted to Intensive Care Units (ICU) in the UK. One of the most common reasons to be admitted to an ICU is the need for respiratory support. Evidence suggests that over 16,500 ICU patients per year (7%) have lung injury of significant severity that proning will be beneficial to improve both oxygenation and chances of survival. Proning describes the technique whereby sedated patients on a ventilator are turned onto their front. Once proned, patients stay on their front for 16-18 hours. Depending upon the patient's condition, this process may be repeated up to five times during an ICU stay, although during the COVID-19 pandemic, some patients were proned up to 10 times. The use of proning has been shown to reduce the risk of death by 17.4%; this is one of the greatest reductions in mortality from a single intervention in intensive care medicine, and this underpins the enthusiasm of clinicians to employ the technique. Whilst proned, a patient's head needs to be turned and their arms repositioned (hereafter termed 'repositioning') regularly to minimise the risk of pressure sores and nerve/organ injuries. This task requires a team of five or more staff and takes 30-60 minutes to perform (more if full Personal Protective Equipment (PPE) is required).

The evidence that proning improves oxygen levels and survival rates in patients who are severely oxygen dependent on ICU is irrefutable. As such, the technique forms an essential component of national and international guidance for ICU clinicians. Complications associated with proning are well described. To mitigate the risk of complications, national guidance recommends repositioning every 2-4 hours. Greater awareness of the benefits of proning following the COVID-19 pandemic, means that the use of the technique may be more readily employed in the post-pandemic era. This increase, in combination with the unwieldy, demanding and far from risk free repositioning process (described below), means there is an urgent need to explore safer and more efficient repositioning techniques.

Repositioning is currently carried out in one of four ways:

1. The patient is slid up the bed to allow their supported head (now clear of the mattress) to be rotated before returning to the original position. This is the most common method in the UK and is recommended in national and international guidance. It requires at least 5 staff and is associated with a significant manual handling exercise.
2. A hoist can be used to lift the patient off the bed to allow repositioning whilst elevated. Hoists are large devices that require 3-5 staff to operate, they can be difficult to manoeuvre and are typically limited in number on an ICU. This approach requires the insertion/removal of slings, takes approximately the same amount of time as a manual turn described above, and can lead to unpredictable movement of the patient whilst suspended.
3. A specialist proning bed can be used. This is prohibitively expensive (£800+ per day), complicated and requires large areas for storage when not in use. This approach requires a specialist bed per patient, thereby limiting the number of patients that can be simultaneously proned on any given ICU. This approach is the least preferred and least used repositioning method.
4. Patients can be lifted by staff on the sheet on which they lie whilst one individual turns the head. This requires at least 5 members of staff and is exceptionally demanding from a manual handling perspective, particularly if patients are obese.

Repositioning is a labour-intensive task for staff on ICU but remains essential for patients. Over 1 million ICU staff hours are required in the UK each year for repositioning. This phenomenal staff drain has consequences for ICUs and is associated with several risks:

At least 5 staff are required to reposition the patient every 2-4 hours. This mandates drawing staff from across the ICU and leads to nurses having to leave other patients to support the repositioning exercise. This results in recurrent interruptions in care for other patients who are critically dependent on the drugs or machines which the nurses oversee. This practice necessitates breaches of national standards on nurse:patient ratios and jeopardises the lives of other patients.

Any adverse event of an unsupervised patient on ICU would be all but impossible to defend medico-legally; liberating nurses to care for their own patients is therefore vital.

Staff shortages on ICU in the post-pandemic era may be more significant than they were pre-pandemic, exacerbating the challenges of liberating staff to perform repositioning.

The process of repositioning is currently far from risk free. As sedated, ventilated patients are moved about the bed, there is a risk of removal or displacement of lines or tubes on which the patient's life is continually and critically dependent. This occurs in up to 12.5% of proned patients.

Improper repositioning risks damage to organs such as the eyes, liver, pancreas or genitals and exposes patients to pressure sores, which are the most common source of litigation of ICUs in the UK.

Recurrent repositioning is manually demanding for staff. Manual handling injuries cost the NHS £18bn in 2019/2020, and any device which reduces this risk will ease staffing problems and the fiscal burden on the NHS as a whole.

Staff burnout remains an ongoing challenge on ICU, deepening the staffing crisis. A device which unburdens staff will reduce burnout and staffing challenges.

The researchers have developed an Inflatable Prone Repositioning Device (IPRD) known as the 'BathMat' that improves the safety and ease of repositioning patients while reducing the number of staff and the time required. The BathMat consists of a multi-vessel inflatable pillow, placed underneath a proned patient, which can be inflated to raise the patient's chest and hips. With the patient raised, repositioning of the head and arms can occur with ease, before the device is deflated and the patient is returned to the resting position. The BathMat has four main benefits for patients and staff:

1. Repositioning of the head and arms occurs without the risks described above.
2. It reduces the number of staff required from 5 to 2.
3. It reduces the time it takes for repositioning from 30-60 minutes to 10 minutes.
4. It removes the majority of the manual handling workload.

This study is required to demonstrate the effectiveness of this device in the clinical setting, and provide data regarding its safety, useability and reliability.

This is a randomised, multicentre, single blind crossover study of repositioning in ventilated proned patients using the BathMat vs conventional care across four Intensive Care Units in England. The researchers aim to recruit 30 patients over 12 months of recruitment. This is sufficient to detect a decrease in repositioning time of at least 10 minutes with a power of over 95%.

ELIGIBILITY:
Inclusion Criteria: Any sedated, ventilated patient over 18 years of age identified as requiring proning by a senior ICU clinician.

Exclusion Criteria:

Patients who are:

* Awake
* Pregnant
* Under guardianship
* In their first proning session in the current ICU admission who have already been repositioned 2 or more times using standard care prior to recruitment to the study.
* Over 200 kg
* Under 150cm and over 205cm
* Patients who have already been proned using conventional methods in the current ICU admission
* Patients who have broken skin on the anterior chest or abdominal wall

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Time taken to reposition | From enrollment until proning no longer clinically indicated, an average of 60 hours.
  Time taken from the time the first assistant arrives at the bedside to reposition until the repositioning exercise is completed.

SECONDARY OUTCOMES:
Assessment of the number of repositioning exercises undertaken for each patient within a proning intervention. | From enrollment until proning no longer clinically indicated, an average of 60 hours.
  The total number of repositioning exercises performed per proning session
The number of minor or major adverse incidents associated with repositioning patients whilst in the prone position. This includes events such as line or tube displacement. | From enrollment until proning no longer clinically indicated, an average of 60 hours.
  Number of complications associated with proning in each study arm
The manual handling requirement to reposition | From enrollment until proning no longer clinically indicated, an average of 60 hours.
  The difference in perceived effort of repositioning between standard care and when using the BathMat as measured by likert scale of effort required by bedside nurse.
In patients who suffered a major or minor adverse event (as defined in secondary outcome b), assessment of the healthcare costs relating to that event at 3 months following ICU discharge. | 3 months from enrollment
  The health economic cost of complications of proning

CONTACTS AND LOCATIONS:
Locations (1):
- North Bristol Trust, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Only IPD collected for the results of the trial will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: March 2025-June 2026
Access Criteria: IPD and supporting information will be available once published

REFERENCES:
- [Derived] Condry J, Georgiou A, Vangsgaard A, Mills H, Smith T, Hunt A, Lunt AJG. A randomised crossover trial of staff time with proned patients in the ICU using the 'BathMat'. Trials. 2025 Nov 13;26(1):503. doi: 10.1186/s13063-025-09221-x. PMID 41233869